CLINICAL TRIAL: NCT02362503
Title: A Multi-arm, Phase 3, Randomized, Placebo Controlled, Double Blind Clinical Trial to Investigate the Efficacy and Safety of Fostemsavir (BMS-663068/GSK3684934) in Heavily Treatment Experienced Subjects Infected With Multi-drug Resistant HIV-1 (BRIGHTE Study)
Brief Title: Attachment Inhibitor Comparison in Heavily Treatment Experienced Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 205888; AI438-047 (Other: Bristol-Myers Squibb); 2014-002111-41 (EudraCT Number)
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — fostemsavir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A1: BMS-663068 (Experimental): Phase 1: BMS-663068 600 mg tablets orally twice daily for 8 days. Phase 2: BMS-663068 600 mg tablets orally twice daily for 48 weeks or longer.
  Interventions: Drug: BMS-663068
- B1: Placebo + BMS-663068 (Active Comparator): Phase 1: Placebo twice daily for 8 days. Phase 2: BMS-663068 600 mg tablets orally twice daily for 48 weeks or longer.
  Interventions: Drug: BMS-663068; Other: Placebo
- BMS-663068 (Experimental): BMS-663068 600 mg tablets orally twice daily for 48 weeks or longer.
  Interventions: Drug: BMS-663068

INTERVENTIONS:
Drug: BMS-663068 — BMS-663068
Other: Placebo — Placebo
  Arms: B1: Placebo + BMS-663068

SUMMARY:
The purpose of this study is to determine whether the BMS Attachment Inhibitor (BMS-663068) is effective in the treatment of heavily treatment experienced HIV-1 patients with multi-drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women with chronic HIV-1 infection
* Antiretroviral-experienced with documented historical or baseline resistance, intolerability, and/or contraindications to antiretrovirals in at least three classes
* Failing current antiretroviral regimen with a confirmed plasma HIV-1 RNA ≥ 400 c/mL (first value from Investigator, second from Screening labs)
* Must have ≤ 2 classes with at least 1 but no more than 2 fully-active antiretrovirals remaining which can be effectively combined to form a viable new regimen, based on current and/or documented historical resistance testing and tolerability and safety
* Able to receive ≥ 1 fully active approved antiretroviral as part of the OBT from Day 9 onwards in the Randomized Cohort
* Subjects without any remaining fully active approved antiretroviral may be enrolled in the Non-Randomized Cohort

Exclusion Criteria:

* Chronic untreated Hepatitis B virus (HBV) (however, patients with chronic treated HBV are eligible)
* HIV-2 infection
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 7 x ULN
* Alkaline Phosphatase > 5 x ULN
* Bilirubin ≥ 1.5 x Upper limit of normal (ULN) (unless subject is currently on atazanavir and has predominantly unconjugated hyperbilirubinemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2026-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (105):
- United States (30):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Wilton Manors, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
- Argentina (5):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Rosario
- Australia (2):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Melbourne, Victoria
- Belgium (2):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
- Brazil (8):
  - GSK Investigational Site, Belo Horizonte
  - GSK Investigational Site, Campinas
  - GSK Investigational Site, Curitiba
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, RibeirAo PretoSP
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São Paulo
- Canada (5):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- Chile (2):
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Temuco
- Colombia (2):
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Cali
- France (4):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
- Germany (5):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Dortmund
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Freiburg im Breisgau
  - GSK Investigational Site, München
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki
- GSK Investigational Site, Dublin, Ireland
- Italy (5):
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Monza MB
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Torino
- Mexico (5):
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Distrito Federal
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- GSK Investigational Site, Utrecht, Netherlands
- Peru (2):
  - GSK Investigational Site, Iquitos
  - GSK Investigational Site, Lima
- Poland (2):
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
- GSK Investigational Site, Lisbon, Portugal
- GSK Investigational Site, San Juan, Puerto Rico
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Constanța
- Russia (2):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Krasnodar
- South Africa (8):
  - GSK Investigational Site, Auckland Park Johannesb
  - GSK Investigational Site, Benoni
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Observatory Cape Town
  - GSK Investigational Site, Port Elizabeth
- Spain (4):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville
- GSK Investigational Site, Taipei, Taiwan
- United Kingdom (3):
  - GSK Investigational Site, Bournemouth
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, London

REFERENCES:
- [Background] Kozal M, Aberg J, Pialoux G, Cahn P, Thompson M, Molina JM, Grinsztejn B, Diaz R, Castagna A, Kumar P, Latiff G, DeJesus E, Gummel M, Gartland M, Pierce A, Ackerman P, Llamoso C, Lataillade M; BRIGHTE Trial Team. Fostemsavir in Adults with Multidrug-Resistant HIV-1 Infection. N Engl J Med. 2020 Mar 26;382(13):1232-1243. doi: 10.1056/NEJMoa1902493. PMID 32212519
- [Derived] Benlarbi M, Richard J, Clemente T, Bourassa C, Tolbert WD, Prakash M, Chandravanshi M, Clark A, Pazgier M, Durand M, Castagna A, Finzi A. Fostemsavir Decreases the Levels of Anti-gp120 CD4-Induced Antibodies in Heavily Treatment-Experienced People With HIV. J Infect Dis. 2025 Sep 24:jiaf461. doi: 10.1093/infdis/jiaf461. Online ahead of print. PMID 40990223
- [Derived] Clark A, Prakash M, Chabria S, Pierce A, Castillo-Mancilla JR, Wang M, Du F, Tenorio AR. Inflammatory Biomarker Reduction With Fostemsavir Over 96 Weeks in Heavily Treatment-Experienced Adults With Multidrug-Resistant HIV-1 in the BRIGHTE Study. Open Forum Infect Dis. 2024 Aug 26;11(9):ofae469. doi: 10.1093/ofid/ofae469. eCollection 2024 Sep. PMID 39233711
- [Derived] Llibre JM, Aberg JA, Walmsley S, Velez J, Zala C, Crabtree Ramirez B, Shepherd B, Shah R, Clark A, Tenorio AR, Pierce A, Du F, Li B, Wang M, Chabria S, Warwick-Sanders M. Long-term safety and impact of immune recovery in heavily treatment-experienced adults receiving fostemsavir for up to 5 years in the phase 3 BRIGHTE study. Front Immunol. 2024 May 28;15:1394644. doi: 10.3389/fimmu.2024.1394644. eCollection 2024. PMID 38863717
- [Derived] Aberg JA, Shepherd B, Wang M, Madruga JV, Mendo Urbina F, Katlama C, Schrader S, Eron JJ, Kumar PN, Sprinz E, Gartland M, Chabria S, Clark A, Pierce A, Lataillade M, Tenorio AR. Week 240 Efficacy and Safety of Fostemsavir Plus Optimized Background Therapy in Heavily Treatment-Experienced Adults with HIV-1. Infect Dis Ther. 2023 Sep;12(9):2321-2335. doi: 10.1007/s40121-023-00870-6. Epub 2023 Sep 26. PMID 37751019
- [Derived] Gartland M, Cahn P, DeJesus E, Diaz RS, Grossberg R, Kozal M, Kumar P, Molina JM, Mendo Urbina F, Wang M, Du F, Chabria S, Clark A, Garside L, Krystal M, Mannino F, Pierce A, Ackerman P, Lataillade M. Week 96 Genotypic and Phenotypic Results of the Fostemsavir Phase 3 BRIGHTE Study in Heavily Treatment-Experienced Adults Living with Multidrug-Resistant HIV-1. Antimicrob Agents Chemother. 2022 Jun 21;66(6):e0175121. doi: 10.1128/aac.01751-21. Epub 2022 May 3. PMID 35502922
- [Derived] Anderson SJ, Murray M, Cella D, Grossberg R, Hagins D, Towner W, Wang M, Clark A, Pierce A, Llamoso C, Ackerman P, Lataillade M. Patient-Reported Outcomes in the Phase III BRIGHTE Trial of the HIV-1 Attachment Inhibitor Prodrug Fostemsavir in Heavily Treatment-Experienced Individuals. Patient. 2022 Jan;15(1):131-143. doi: 10.1007/s40271-021-00534-y. Epub 2021 Jun 28. PMID 34180035
- [Derived] Lataillade M, Lalezari JP, Kozal M, Aberg JA, Pialoux G, Cahn P, Thompson M, Molina JM, Moreno S, Grinsztejn B, Diaz RS, Castagna A, Kumar PN, Latiff GH, De Jesus E, Wang M, Chabria S, Gartland M, Pierce A, Ackerman P, Llamoso C. Safety and efficacy of the HIV-1 attachment inhibitor prodrug fostemsavir in heavily treatment-experienced individuals: week 96 results of the phase 3 BRIGHTE study. Lancet HIV. 2020 Nov;7(11):e740-e751. doi: 10.1016/S2352-3018(20)30240-X. PMID 33128903
- [Derived] Lagishetty C, Moore K, Ackerman P, Llamoso C, Magee M. Effects of Temsavir, Active Moiety of Antiretroviral Agent Fostemsavir, on QT Interval: Results From a Phase I Study and an Exposure-Response Analysis. Clin Transl Sci. 2020 Jul;13(4):769-776. doi: 10.1111/cts.12763. Epub 2020 Mar 19. PMID 32027457

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2 cohort Phase 3 study conducted in heavily treatment experienced (HTE) participants infected with multi-drug resistant human immunodeficiency virus (HIV)-1. Participants were assigned to either the Randomized Cohort (participants received either fostemsavir or placebo) or Non-randomized Cohort (all participants received fostemsavir).
Pre-assignment Details: A total of 731 participants were screened, of which 371 were included in either Randomized Cohort or Non-randomized Cohort and received at least one dose of study treatment. The results presented are based on Week 96 interim analysis. Data collection is still on-going and additional results will be provided after study completion.
Groups:
- Randomized Cohort-Placebo: Eligible participants in the Randomized Cohort had one to two fully active antiretrovirals remaining at Baseline. Participants received placebo twice daily (BID) along with their currently failing antiretroviral regimen for 8 days during the randomized, double-blind period. During the open-label period, all participants received fostemsavir 600 mg BID with an optimized background therapy (OBT).
- Randomized Cohort-fostemsavir 600 mg BID: Eligible participants in the Randomized Cohort had one to two fully active antiretrovirals remaining at Baseline. Participants received fostemsavir 600 milligram (mg) BID along with currently failing antiretroviral regimen for 8 days during the randomized, double-blind period. During the open-label period, all participants continued to receive fostemsavir 600 mg BID with an OBT.
- Non-randomized Cohort-fostemsavir 600 mg BID-Open Label Period: Eligible participants in the Non-randomized Cohort had zero remaining fully active and approved antiretroviral regimens at Baseline. Participants received fostemsavir 600 mg BID in combination with OBT.
Period: Double-blind Period-Up to 8 Days
Arm/Group | Randomized Cohort-Placebo | Randomized Cohort-fostemsavir 600 mg BID | Non-randomized Cohort-fostemsavir 600 mg BID-Open Label Period
Started | 69 | 203 | 0
Completed | 68 | 199 | 0
Not Completed | 1 | 4 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — No longer meets study criteria | 0 | 1 | 0
Period: Open Label Period-Up to 96 Weeks
Arm/Group | Randomized Cohort-Placebo | Randomized Cohort-fostemsavir 600 mg BID | Non-randomized Cohort-fostemsavir 600 mg BID-Open Label Period
Started | 68 | 199 | 99
Completed | 0 | 0 | 0
Not Completed | 68 | 199 | 99
Not completed — Other | 0 | 1 | 1
Not completed — No longer meets criteria | 0 | 4 | 4
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Non-compliance with study drug | 3 | 8 | 6
Not completed — Lost to Follow-up | 4 | 3 | 1
Not completed — Death | 1 | 7 | 15
Not completed — Withdrawal by Subject | 0 | 5 | 1
Not completed — Adverse Event | 3 | 2 | 4
Not completed — Lack of Efficacy | 3 | 9 | 6
Not completed — Ongoing at the time of analysis | 54 | 159 | 61

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Cohort-Placebo | Randomized Cohort-fostemsavir 600 mg BID | Non-randomized Cohort-fostemsavir 600 mg BID-Open Label Period | Total
Number analyzed (Participants) | 69 | 203 | 99 | 371
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (11.02) | 45.2 (12.72) | 48.1 (11.53) | 45.6 (12.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 60 | 10 | 82
  Male | 57 | 143 | 89 | 289
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race customized: Black or African American | 18 | 42 | 23 | 83
  Race customized: American Indian or Alaska Native | 1 | 6 | 1 | 8
  Race customized: Asian | 0 | 2 | 0 | 2
  Race customized: Native Hawaiian or other Pacific islander | 0 | 1 | 0 | 1
  Race customized: White | 48 | 137 | 74 | 259
  Race customized: Mixed | 1 | 6 | 1 | 8
  Race customized: Hispanic | 0 | 2 | 0 | 2
  Race customized: Mestizo | 1 | 2 | 0 | 3
  Race customized: North African | 0 | 1 | 0 | 1
  Race customized: Mulatto | 0 | 1 | 0 | 1
  Race customized: Brown | 0 | 2 | 0 | 2
  Race customized: White and African descent | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Logarithm to the Base 10 (log10) HIV-1 Ribonucleic Acid (RNA) From Day 1 at Day 8-Randomized Cohort
Description: Plasma samples were collected for analysis of HIV-1 RNA. Mean change in log10 HIV-1 RNA from Day 1 was estimated using analysis of covariance (ANCOVA) with log10 HIV-1 RNA change from Day 1 at Day 8 as dependent variable, treatment (fostemsavir or placebo) as an independent variable, and Day 1 log10 HIV-1 RNA as a continuous covariate. Change from Day 1 was calculated as value at Day 8 minus value at Day 1. The analysis was performed on Intent-to-Treat Exposed (ITT-E) Population which comprised of all randomized participants who received at least one dose of study treatment. Missing HIV-1 RNA values at Day 8 were imputed using (a) Day 1 Observation Carried Forward (D1OCF) for participants without a value during blinded treatment (i.e, imputing a zero change from Day 1) or (b) Last Observation Carried Forward (LOCF) for participants with an early value during blinded treatment before the Day 8 analysis visit window.
Time Frame: Day 1 and Day 8
Population: ITT-E Population. Participants with missing Day 1 HIV-1 RNA values were not analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Log10 copies per milliliter (c/mL)
Arm/Group | Randomized Cohort-Placebo | Randomized Cohort-fostemsavir 600 mg BID
Number analyzed (Participants) | 69 | 201
Log10 copies per milliliter (c/mL) | -0.166 [-0.326 to -0.007] | -0.791 [-0.885 to -0.698]
Statistical Analysis 1: Comparison: Randomized Cohort-Placebo vs Randomized Cohort-fostemsavir 600 mg BID; Test type: Superiority; p < 0.0001, ANCOVA — Hypothesis test:µfostemsavir=µPlacebo where µ is a common intercept; Mean Difference (Net) = -0.625, 95% CI 2-sided [-0.810 to -0.441] — Difference in covariate-adjusted least squares means between treatment groups (Fostemsavir 600 mg BID-Placebo) is presented

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA Decreases From Day 1 That Exceed 0.5 log10 c/mL and 1.0 log10 c/mL at Day 8-Randomized Cohort
Description: The percentage of participants in the Randomized Cohort with HIV-1 RNA decreases from Day 1 that exceed 0.5 log10 c/mL and 1.0 log10 c/mL at Day 8 was determined by comparing HIV-1 RNA Day 1 measurement of each participant to their Day 8 measurement. This was an ITT analysis that classified participants without HIV-1 RNA at Day 1 or Day 8 as failures. The percentage of responders along with 95% confidence interval based on Wilson score is presented.
Time Frame: Day 1 and Day 8
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Randomized Cohort-Placebo | Randomized Cohort-fostemsavir 600 mg BID
Number analyzed (Participants) | 69 | 203
Percentage of participants
  >0.5 log10 c/mL | 18.84 [11.35 to 29.61] | 64.53 [57.74 to 70.79]
  >1.0 log10 c/mL | 10.14 [5.00 to 19.49] | 45.81 [39.10 to 52.68]
Statistical Analysis 1: Comparison: Randomized Cohort-Placebo vs Randomized Cohort-fostemsavir 600 mg BID; Test type: Other; Mean Difference (Net) = 45.69, 95% CI 2-sided [32.95 to 55.45] — Difference between treatment groups (fostemsavir 600 mg BID-Placebo) and 95% confidence interval using Newcombe method is presented for >0.5 log10 c/mL
Statistical Analysis 2: Comparison: Randomized Cohort-Placebo vs Randomized Cohort-fostemsavir 600 mg BID; Test type: Other; Mean Difference (Net) = 35.67, 95% CI 2-sided [24.16 to 44.25] — Difference between treatment groups (fostemsavir 600 mg BID-Placebo) and 95% confidence interval using Newcombe method is presented for >1.0 log10 c/mL

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA <40 c/mL at Weeks 24, 48 and 96-Randomized Cohort
Description: The durability of response (that is, the number of participants achieving HIV-1 RNA <40 c/mL) at Weeks 24, 48 and 96 of open-label fostemsavir plus OBT in the Randomized Cohort was assessed using the Food and Drug Administration (FDA) snapshot algorithm in which participants without HIV-1 RNA at Weeks 24, 48 and 96 or those who changed OBT due to lack of efficacy through Weeks 24, 48 and 96 were counted as failures. The percentage of participants in the Randomized Cohort who achieved virologic success (HIV-1 RNA <40 c/mL) at Weeks 24, 48 and 96 is presented along with 95% Wilson confidence interval. All the participants received fostemsavir during the open-label period irrespective of the original arms to which they were randomized; hence, the combined totals for Randomized Cohort is presented as pre-specified in protocol and reporting and analysis plan.
Time Frame: At Weeks 24, 48 and 96
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Randomized Cohort: Eligible participants in the Randomized Cohort had one to two fully active antiretrovirals remaining at Baseline. Participants were randomized to receive fostemsavir 600 mg BID or placebo along with their current failing antiretroviral regimen during the double-blind period for 8 days. During the open-label period, all participants received open-label fostemsavir 600 mg BID in combination with OBT for at least 96 weeks.
Arm/Group | Randomized Cohort
Number analyzed (Participants) | 272
Percentage of participants
  Week 24 | 53 [47.0 to 58.8]
  Week 48 | 54 [47.7 to 59.5]
  Week 96 | 60 [54.0 to 65.6]

4. Secondary Outcome: Number of Participants With On-treatment Serious Adverse Events (SAEs) and Adverse Events (AEs) Leading to Discontinuation (AELD)-Randomized Cohort
Description: An SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or causes prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; an important medical event that may jeopardize the participant or require intervention. Number of participants with on-treatment SAEs and AEs leading to withdrawal of study treatment is presented. SAEs and AELDs were collected in Safety Population which comprised of all participants who received at least one dose of study treatment. All the participants received fostemsavir during the open-label period irrespective of the original arms to which they were randomized; hence, the combined totals for Randomized Cohort is presented as pre-specified in protocol and reporting and analysis plan.
Time Frame: Up to Week 96 analysis cut-off date
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Cohort
Number analyzed (Participants) | 272
Participants
  SAE | 92
  AELD | 14

5. Secondary Outcome: Number of Participants With Toxicity Grade Increase in Clinical Chemistry Results to Grade 3-4 Relative to Baseline-Randomized Cohort
Description: Laboratory toxicities were graded for severity according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) grading system: Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe); Grade 4 (potentially life-threatening). Baseline is defined as the latest pre-dose assessment. The number of participants with clinical chemistry toxicity grade increase to Grade 3-4 at anytime post-Baseline relative to Baseline is presented. All the participants received fostemsavir during the open-label period irrespective of the original arms to which they were randomized; hence, the combined totals for Randomized Cohort is presented as pre-specified in protocol and reporting and analysis plan.
Time Frame: Baseline and up to Week 96 analysis cut-off date
Population: Safety Population. Only participants with data available at the specified time points were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Cohort
Number analyzed (Participants) | 272
Participants
  Albumin; n=268: number analyzed (Participants) | 268
  Albumin; n=268 | 1
  Alkaline phosphatase; n=268: number analyzed (Participants) | 268
  Alkaline phosphatase; n=268 | 3
  Alanine aminotransferase; n=268: number analyzed (Participants) | 268
  Alanine aminotransferase; n=268 | 14
  Amylase; n=268: number analyzed (Participants) | 268
  Amylase; n=268 | 2
  Aspartate aminotransferase; n=268: number analyzed (Participants) | 268
  Aspartate aminotransferase; n=268 | 10
  Bicarbonate; n=268: number analyzed (Participants) | 268
  Bicarbonate; n=268 | 1
  Direct bilirubin; n=268: number analyzed (Participants) | 268
  Direct bilirubin; n=268 | 20
  Bilirubin; n=268: number analyzed (Participants) | 268
  Bilirubin; n=268 | 7
  Calcium; n=268: number analyzed (Participants) | 268
  Calcium; n=268 | 9
  Cholesterol; n=221: number analyzed (Participants) | 221
  Cholesterol; n=221 | 10
  Creatine kinase; n=268: number analyzed (Participants) | 268
  Creatine kinase; n=268 | 6
  Creatinine; n=268: number analyzed (Participants) | 268
  Creatinine; n=268 | 52
  Estimated creatinine clearance; n=268: number analyzed (Participants) | 268
  Estimated creatinine clearance; n=268 | 75
  Glucose/hyperglycemia; n=267: number analyzed (Participants) | 267
  Glucose/hyperglycemia; n=267 | 6
  Glucose/hypoglycemia; n=267: number analyzed (Participants) | 267
  Glucose/hypoglycemia; n=267 | 2
  Potassium/hyperkalemia; n=268: number analyzed (Participants) | 268
  Potassium/hyperkalemia; n=268 | 4
  Potassium/hypokalemia; n=268: number analyzed (Participants) | 268
  Potassium/hypokalemia; n=268 | 0
  Low density lipoprotein (LDL) cholesterol; n=216: number analyzed (Participants) | 216
  Low density lipoprotein (LDL) cholesterol; n=216 | 8
  Lipase; n=268: number analyzed (Participants) | 268
  Lipase; n=268 | 13
  Sodium/hypernatremia; n=268: number analyzed (Participants) | 268
  Sodium/hypernatremia; n=268 | 0
  Sodium/hyponatremia; n=268: number analyzed (Participants) | 268
  Sodium/hyponatremia; n=268 | 0
  Triglycerides; n=221: number analyzed (Participants) | 221
  Triglycerides; n=221 | 11
  Urate; n=268: number analyzed (Participants) | 268
  Urate; n=268 | 9

6. Secondary Outcome: Number of Participants With Toxicity Grade Increase in Hematology Results to Grade 3-4 Relative to Baseline-Randomized Cohort
Description: Laboratory toxicities were graded for severity according to the DAIDS grading system: Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe); Grade 4 (potentially life-threatening). Baseline is defined as the latest pre-dose assessment. The number of participants with hematology toxicity grade increase to Grade 3-4 at anytime post-Baseline relative to Baseline is presented. All the participants received fostemsavir during the open-label period irrespective of the original arms to which they were randomized; hence, the combined totals for Randomized Cohort is presented as pre-specified in protocol and reporting and analysis plan.
Time Frame: Baseline and up to Week 96 analysis cut-off date
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Cohort
Number analyzed (Participants) | 272
Participants
  Hemoglobin; n=268: number analyzed (Participants) | 268
  Hemoglobin; n=268 | 16
  Neutrophils; n=268: number analyzed (Participants) | 268
  Neutrophils; n=268 | 10
  Platelets; n=267: number analyzed (Participants) | 267
  Platelets; n=267 | 2
  Leukocytes; n=268: number analyzed (Participants) | 268
  Leukocytes; n=268 | 4

7. Secondary Outcome: Number of Participants With Centers for Disease Control (CDC) Class C Events-Randomized Cohort
Description: Disease progression during open label fostemsavir plus OBT was assessed based on the occurrence of new AIDS defining events (CDC Class C events) or death. The number of participants with on-treatment CDC Class C AIDS events is presented. All the participants received fostemsavir during the open-label period irrespective of the original arms to which they were randomized; hence, the combined totals for Randomized Cohort is presented as pre-specified in protocol and reporting and analysis plan.
Time Frame: Up to Week 96 analysis cut-off date
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Cohort
Number analyzed (Participants) | 272
Participants | 23

8. Secondary Outcome: Change From Day 1 in Cluster of Differentiation (CD) 4+ T-cell Count at Day 8-Randomized Cohort
Description: CD4+ T- cell counts were assessed by flow cytometry. Mean change in CD4+ T- cell count from Day 1 at Day 8 was analyzed using one-way ANCOVA with change of CD4+ cell counts from Day 1 at Day 8 as the dependent variable, treatment (fostemsavir or placebo) as an in-dependent variable, and Day 1 CD4+ cell count as a continuous covariate. Change from Day 1 was calculated as value at Day 8 minus value at Day 1. Missing CD4+ cell count values at Day 8 were imputed using (a) D1OCF for participants without a value during blinded treatment (i.e., imputing a zero change from Day 1), or (b) LOCF for participants with an early value during blinded treatment before the Day 8 analysis visit window.
Time Frame: Day 1 and Day 8
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Cells per cubic millimeter
Arm/Group | Randomized Cohort-Placebo | Randomized Cohort-fostemsavir 600 mg BID
Number analyzed (Participants) | 69 | 196
Cells per cubic millimeter | 18.9 [4.7 to 33.0] | 18.5 [10.1 to 26.8]
Statistical Analysis 1: Comparison: Randomized Cohort-Placebo vs Randomized Cohort-fostemsavir 600 mg BID; Test type: Other; Mean Difference (Net) = -0.4, 95% CI 2-sided [-16.8 to 16.0] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change in CD4+ T- Cell Count Percentage From Day 1 at Day 8-Randomized Cohort
Description: CD4+ T- cell counts were assessed by flow cytometry. Mean change in CD4+ T- cell count percentage from Day 1 at Day 8 was analyzed using one-way ANCOVA with change of CD4+ cell count percentage from Day 1 at Day 8 as the dependent variable, treatment (fostemsavir or placebo) as an independent variable, and Day 1 CD4+ cell count percentage as a continuous covariate. Change from Day 1 was calculated as value at Day 8 minus value at Day 1. Missing CD4+ cell count values at Day 8 were imputed using (a) D1OCF for participants without a value during blinded treatment (ie, imputing a zero change from Day 1), or (b) LOCF for participants with an early value during blinded treatment before the Day 8 analysis visit window.
Time Frame: Day 1 and Day 8
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of CD4+T- cells
Arm/Group | Randomized Cohort-Placebo | Randomized Cohort-fostemsavir 600 mg BID
Number analyzed (Participants) | 69 | 196
Percentage of CD4+T- cells | 0.243 [-0.216 to 0.703] | 0.860 [0.588 to 1.133]
Statistical Analysis 1: Comparison: Randomized Cohort-Placebo vs Randomized Cohort-fostemsavir 600 mg BID; Test type: Other; Mean Difference (Net) = 0.617, 95% CI 2-sided [0.082 to 1.151] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change From Baseline in log10 HIV-1 RNA for Fostemsavir When Given With OBT Through Week 96-Randomized Cohort
Description: Blood samples were collected for the analysis of HIV-1 RNA. Baseline is defined as the last non-missing value on or before the date of first dose of study treatment. Change from Baseline was calculated as the value at post-dose visit minus the value at Baseline. All the participants received fostemsavir during the open-label period irrespective of the original arms to which they were randomized; hence, the combined totals for Randomized Cohort is presented as pre-specified in protocol and reporting and analysis plan.
Time Frame: Baseline and at Day 8, Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84 and 96
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Log10 c/mL
Arm/Group | Randomized Cohort
Number analyzed (Participants) | 272
Log10 c/mL
  Day 8; n=262: number analyzed (Participants) | 262
  Day 8; n=262 | -0.656 (0.7536)
  Week 4; n=262: number analyzed (Participants) | 262
  Week 4; n=262 | -2.051 (1.0717)
  Week 8; n=256: number analyzed (Participants) | 256
  Week 8; n=256 | -2.207 (1.1416)
  Week 12; n=248: number analyzed (Participants) | 248
  Week 12; n=248 | -2.237 (1.2105)
  Week 16; n=249: number analyzed (Participants) | 249
  Week 16; n=249 | -2.277 (1.2834)
  Week 24; n=246: number analyzed (Participants) | 246
  Week 24; n=246 | -2.297 (1.2788)
  Week 36; n=238: number analyzed (Participants) | 238
  Week 36; n=238 | -2.332 (1.2265)
  Week 48; n=233: number analyzed (Participants) | 233
  Week 48; n=233 | -2.324 (1.2876)
  Week 60; n=223: number analyzed (Participants) | 223
  Week 60; n=223 | -2.419 (1.1973)
  Week 72; n=221: number analyzed (Participants) | 221
  Week 72; n=221 | -2.427 (1.1542)
  Week 84; n=215: number analyzed (Participants) | 215
  Week 84; n=215 | -2.455 (1.1930)
  Week 96; n=214: number analyzed (Participants) | 214
  Week 96; n=214 | -2.476 (1.1984)

11. Secondary Outcome: Change From Baseline in CD4+ T- Cell Count Through Week 96-Randomized Cohort
Description: CD4+ T- cell counts were assessed by flow cytometry. Baseline is defined as the last non-missing value on or before the date of first dose of study treatment. Change from Baseline was calculated as the value at post-dose visit minus the value at Baseline.
Time Frame: Baseline and at Day 8, Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | Randomized Cohort
Number analyzed (Participants) | 272
Cells per cubic millimeter
  Day 8; n=255: number analyzed (Participants) | 255
  Day 8; n=255 | 19.8 (60.98)
  Week 4; n=259: number analyzed (Participants) | 259
  Week 4; n=259 | 48.9 (131.75)
  Week 8; n=254: number analyzed (Participants) | 254
  Week 8; n=254 | 61.5 (113.47)
  Week 12; n=249: number analyzed (Participants) | 249
  Week 12; n=249 | 79.0 (123.31)
  Week 16; n=245: number analyzed (Participants) | 245
  Week 16; n=245 | 84.1 (107.26)
  Week 24; n=247: number analyzed (Participants) | 247
  Week 24; n=247 | 90.4 (112.10)
  Week 36; n=234: number analyzed (Participants) | 234
  Week 36; n=234 | 109.7 (119.50)
  Week 48; n=228: number analyzed (Participants) | 228
  Week 48; n=228 | 138.9 (135.06)
  Week 60; n=215: number analyzed (Participants) | 215
  Week 60; n=215 | 162.9 (157.69)
  Week 72; n=217: number analyzed (Participants) | 217
  Week 72; n=217 | 172.1 (184.81)
  Week 84; n=203: number analyzed (Participants) | 203
  Week 84; n=203 | 190.8 (165.63)
  Week 96; n=213: number analyzed (Participants) | 213
  Week 96; n=213 | 204.7 (191.28)

12. Secondary Outcome: Change From Baseline in CD4+ T- Cell Count Percentage Through Week 96
Description: Percentage CD4+ T- cell counts were assessed by flow cytometry. Baseline is defined as the last non-missing value on or before the date of first dose of study treatment. Change from Baseline was calculated as the value at post-dose visit minus the value at Baseline.
Time Frame: Baseline and at Day 8, Weeks 4, 8, 12, 16, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of CD4+ T- cells
Groups:
- Randomized Cohort: Eligible participants in the Randomized Cohort had one to two fully active antiretrovirals remaining at Baseline. Participants were randomized to receive fostemsavir 600 mg or placebo along with their current failing antiretroviral regimen during the double-blind period for 8 days. During the open-label period, all participants received open-label fostemsavir 600 mg BID in combination with OBT for at least 96 weeks
Arm/Group | Randomized Cohort
Number analyzed (Participants) | 272
Percentage of CD4+ T- cells
  Day 8; n=255: number analyzed (Participants) | 255
  Day 8; n=255 | 0.75 (1.970)
  Week 4; n=259: number analyzed (Participants) | 259
  Week 4; n=259 | 2.30 (4.643)
  Week 8; n=254: number analyzed (Participants) | 254
  Week 8; n=254 | 2.36 (4.392)
  Week 12; n=249: number analyzed (Participants) | 249
  Week 12; n=249 | 3.00 (4.945)
  Week 16; n=245: number analyzed (Participants) | 245
  Week 16; n=245 | 3.51 (4.979)
  Week 24; n=247: number analyzed (Participants) | 247
  Week 24; n=247 | 4.26 (4.828)
  Week 36; n=234: number analyzed (Participants) | 234
  Week 36; n=234 | 5.06 (5.256)
  Week 48; n=228: number analyzed (Participants) | 228
  Week 48; n=228 | 6.51 (5.531)
  Week 60; n=215: number analyzed (Participants) | 215
  Week 60; n=215 | 7.00 (5.940)
  Week 72; n=217: number analyzed (Participants) | 217
  Week 72; n=217 | 7.02 (5.726)
  Week 84; n=203: number analyzed (Participants) | 203
  Week 84; n=203 | 7.68 (5.798)
  Week 96; n=213: number analyzed (Participants) | 213
  Week 96; n=213 | 8.44 (6.409)

13. Secondary Outcome: Number of Participants With Treatment-emergent Viral Genotypic Substitution of Interest in the GP160 Domain as a Measure of Genotypic Resistance-Randomized Cohort
Description: Plasma samples were collected for emergent drug resistance testing. The number of participants with emergent viral genotypic substitutions of interest in the GP160 domain was identified by the next-generation sequencing (NGS) assay. Protocol defined virologic failure (PDVF) through Week 96 Population comprised of all participants with available phenotypic and genotypic resistance data meeting at the time protocol defined virologic failure (PDVF) was met. The criteria for PDVF was a) Confirmed, or last available prior to discontinuation, HIV-1 RNA >=400 c/mL at any time after prior confirmed suppression to <400 c/mL prior to Week 24 or Confirmed, or last available prior to discontinuation, > 1 log10 c/mL increase in HIV-1 RNA at any time above nadir level where nadir is >=40 c/mL prior to Week 24. b) Confirmed, or last available prior to discontinuation, HIV-1 RNA >=400 c/mL at or after Week 24.
Time Frame: Week 96
Population: PDVF through Week 96 Population. Only participants available at the specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Cohort
Number analyzed (Participants) | 50
Participants | 24

14. Secondary Outcome: Number of Participants With Indicated Fold Change Ratio (FCR) Using the Monogram PhenoSense Entry Assay-Randomized Cohort
Description: The phenotypic resistance to a drug is defined in terms of a fold change (FC) in IC50s, i.e., the ratio of the 50% inhibitory concentration (IC50) of the clinical isolate to the IC50 of a reference strain (wild type control). FCR was calculated as FC at PDVF divided by Baseline FC. The number of participants with the indicated change (ratio) in the two values at the time of PDVF is presented. FCR<1 indicates that FC is smaller on-treatment than at Baseline. FCR >3 indicates that on-treatment FC is 3 times greater than it was at Baseline.
Time Frame: Week 96
Population: PDVF through Week 96 Population. Only participants available at the specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Cohort
Number analyzed (Participants) | 53
Participants
  <=1 | 19
  >1 to 3 | 10
  >3 to 10 | 5
  >10 to 100 | 1
  >100 to 3000 | 10
  >3000 | 8

ADVERSE EVENTS:
Time Frame: On-treatment non-SAEs and SAEs were collected from the start of study treatment until Week 96 data cut-off date. The data presented for Randomized Cohort-Placebo and Randomized Cohort-fostemsavir 600 mg BID represent safety events during the double-blind period (Up to Day 8). The safety data presented in the Randomized Cohort-Total, Non-Randomized Cohort-fostemsavir 600 mg BID and Fostemsavir Total columns represent safety events during fostemsavir dosing until the Week 96 data cut-off date.
Description: Non-SAEs and SAEs were collected in the Safety Population which comprised of all participants who received at least one dose of study treatment. One participant was excluded from the Randomized Cohort-Total and Total fostemsavir population as the participant took only placebo and had discontinued during the double-blind period.
Groups:
- Non-randomized Cohort-fostemsavir 600 mg BID: This reporting group includes HTE HIV-1 infected participants who were assigned to the Non-randomized Cohort and received fostemsavir 600 mg BID and OBT. Non-randomized Cohort participants are assigned based on their screening status of having no remaining classes of fully active antiretroviral that can combined in a new drug regimen. The data reported are safety events during fostemsavir dosing until the Week 96 data cut-off date.
- Randomized Cohort-Total: This reporting group includes all participants in the Randomized Cohort. The data reported are safety events during fostemsavir dosing until the Week 96 data cut-off date.
- Total Fostemsavir: This reporting group included all enrolled participants (Randomized Cohort and Non-randomized Cohort) and who received fostemsavir 600 mg during the open-label period. The data reported are safety events during fostemsavir dosing until the Week 96 data cut-off date.
Arm/Group | Randomized Cohort-Placebo | Randomized Cohort-fostemsavir 600 mg BID | Non-randomized Cohort-fostemsavir 600 mg BID | Randomized Cohort-Total | Total Fostemsavir
All-Cause Mortality (participants affected / at risk) | 2/69 | 10/203 | 17/99 | 12/271 | 29/370
Serious Adverse Events (participants affected / at risk) | 2/69 | 4/203 | 48/99 | 92/271 | 140/370
Other Adverse Events (participants affected / at risk) | 16/69 | 45/203 | 92/99 | 214/271 | 306/370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Cohort-Placebo (N=69) | Randomized Cohort-fostemsavir 600 mg BID (N=203) | Non-randomized Cohort-fostemsavir 600 mg BID (N=99) | Randomized Cohort-Total (N=271) | Total Fostemsavir (N=370)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 3 (4) | 12 (15) | 15 (19)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 5 (5) | 8 (9)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 6 (6)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 4 (5)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 4 (6)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (4)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (4)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (4)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
HIV-associated neurocognitive disorder (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hepatitis A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 2 (4)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anogenital dysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anorectal cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood HIV RNA increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Central nervous system immune reconstitution inflammatory response (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Disseminated cytomegaloviral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatitis B reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Histoplasmosis disseminated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Kidney rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Meningitis coccidioides (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Meningoencephalitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mononeuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Open fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prostatic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Reactive gastropathy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Salmonella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Septic rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tuberculosis liver (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Cohort-Placebo (N=69) | Randomized Cohort-fostemsavir 600 mg BID (N=203) | Non-randomized Cohort-fostemsavir 600 mg BID (N=99) | Randomized Cohort-Total (N=271) | Total Fostemsavir (N=370)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 8 (8) | 25 (48) | 60 (84) | 85 (132)
Nausea (Gastrointestinal disorders) | 4 (4) | 14 (14) | 21 (31) | 45 (65) | 66 (96)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 15 (21) | 42 (64) | 57 (85)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 19 (24) | 34 (50) | 53 (74)
Headache (Nervous system disorders) | 5 (5) | 6 (6) | 12 (13) | 36 (53) | 48 (66)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 16 (24) | 30 (42) | 46 (66)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 11 (12) | 33 (45) | 44 (57)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (7) | 34 (45) | 39 (52)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 13 (15) | 26 (31) | 39 (46)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 9 (13) | 29 (48) | 38 (61)
Fatigue (General disorders) | 2 (2) | 3 (3) | 16 (16) | 18 (19) | 34 (35)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 11 (13) | 22 (29) | 33 (42)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 9 (11) | 22 (24) | 31 (35)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 6 (7) | 23 (23) | 29 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 12 (14) | 16 (18) | 28 (32)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (5) | 22 (30) | 27 (35)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 10 (13) | 17 (21) | 27 (34)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 10 (14) | 15 (17) | 25 (31)
Asthenia (General disorders) | 2 (2) | 2 (2) | 12 (13) | 11 (14) | 23 (27)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 5 (5) | 17 (18) | 22 (23)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 18 (20) | 21 (23)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 7 (7) | 14 (16) | 21 (23)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 17 (19) | 19 (21)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 5 (6) | 12 (16) | 17 (22)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 6 (8) | 11 (11) | 17 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 11 (15) | 17 (21)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 11 (12) | 16 (17)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 8 (9) | 6 (7) | 14 (16)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 6 (8) | 8 (8) | 14 (16)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 6 (8) | 8 (8) | 14 (16)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (6) | 5 (6) | 11 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (5) | 6 (6) | 11 (11)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 6 (6) | 11 (11)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 9 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 9 (9)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (6) | 4 (4) | 9 (10)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 5 (6) | 3 (4) | 8 (10)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 7 (7)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (15) | 7 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.